CLINICAL TRIAL: NCT04117243
Title: The Efficacy and Safety of Preoperative Intravenous Tranexamic Acid Versus Sublingual Misoprostol in Reducing Blood Loss During and After Elective Cesarean Section Among High Risk Pregnant Cases.
Brief Title: Tranexamic Acid Versus Sublingual Misoprostol in Reducing Blood Loss During Elective CS in High Risk Cases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, Assistant Professor in obstetrics and gynecology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280391
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Post Partum Hemorrhage
Keywords: tranexamic acid; misoprostol; high risk pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Tranexamic Acid; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tranexamic group (Active Comparator): patients will be given 1 gm (10 ml) TXA (Kapron, Amoun, Egypt) diluted in 20 ml of Glucose 5% (administered as intravenous infusion over 5 minutes, at least 15 minutes prior to skin incision).
  Interventions: Drug: Tranexamic acid
- Misoprostol group (Active Comparator): patients will be given 400 microgram misoprostol (2 tablets - Cytotec, Pfizer, G.D. Searle LLC) sublingually immediately before starting skin incision.
  Interventions: Drug: Misoprostol
- oxytocin only group (Active Comparator): patients will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following the delivery of the baby
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — patients will be given 400 microgram misoprostol (2 tablets - Cytotec, Pfizer, G.D. Searle LLC) sublingually immediately before starting skin incision (n=115)
  Other Names: Cytotec
  Arms: Misoprostol group
Drug: Tranexamic acid — patients will be given 1 gm (10 ml) TXA (Kapron, Amoun, Egypt) diluted in 20 ml of Glucose 5% (administered as intravenous infusion over 5 minutes, at least 15 minutes prior to skin incision) (n=115)
  Other Names: Kapron
  Arms: Tranexamic group
Drug: Oxytocin — patients will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following the delivery of the baby (n=115)
  Other Names: syntocinone
  Arms: oxytocin only group

SUMMARY:
The Efficacy and safety of Preoperative Intravenous Tranexamic acid versus Sublingual misoprostol in reducing blood loss during and after Elective Cesarean section among high risk pregnant cases.

DETAILED DESCRIPTION:
The study will include (345) pregnant women attending for elective cesarean delivery in the Kasr Elaini hospital (faculty of medicine - Cairo university).

All the patients will be subjected to informed written consent, full medical history, clinical examination, obstetric ultrasonography, preoperative laboratory tests On the day of the scheduled surgery, participants will be randomly and equally assigned into three groups. Tranexamic group, Misoprostol group and oxytocin-only group (control group). Randomization will be performed using computer-generated random numbers.

In Tranexamic group (n=115), patients will be given 1 gm (10 ml) Tranexamic acid (Kapron, Amoun, Egypt) diluted in 20 ml of Glucose 5% (administered as intravenous infusion over 5 minutes, at least 15 minutes prior to skin incision).

In Misoprostol group (n=115), 400 microgram misoprostol (2 tablets - Cytotec, Pfizer, G.D. Searle LLC) will be administered sublingually by the patients immediately before starting skin incision.

Following the delivery of the baby, patients in both Tranexamic and Misoprostol groups will additionally receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h).

In oxytocin-only group (n=115), patients will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following the delivery of the baby.

All cesarean sections will be done under spinal anesthesia by the following operative steps: pfannenstiel incision, transverse lower uterine segment incision, immediate cord clamping (< 30 seconds) and the placenta will be removed by controlled cord traction after its spontaneous separation, closure of uterus in 2 layers, closure of anterior abdominal wall in anatomical manner (adequate hemostasis will be ensured in all operative steps).

The number and the difference of weight of operative towels (before and after CS) and amount of blood in suction unit will be recorded.

Fluid monitoring will be performed through rate of infusion and urine output. A complete blood count test will be performed 12 hours after delivery.

Estimated Blood Loss (EBL) will be evaluated as follows:

* The number of operative towels used.
* The difference of weight of operative towels (before and after cs) plus the amount of blood in suction unit (we will calculate 1 gram of weight difference equal to 1 ml blood loss).
* the following formula: EBL= EBV x [(Preoperative hematocrit- Postoperative hematocrit)/ Postoperative hematocrit] Where EBV is estimated blood volume of the patient in mL (equals weight in kg × 85).

The time interval between drug administration and fetal delivery will be recorded together with the neonatal outcome (APGAR at 1 and 5 minutes, NICU admission and neonatal death).

All patients will be followed up following the delivery as regard occurrence of primary postpartum hemorrhage (within the first 24 hours), the need for blood transfusion (within the first 24 hours), misoprostol-related side effects (in the first 6 hours) (i.e. shivering, pyrexia >38 C, headache, nausea, vomiting with or without the need for antiemetic drugs) and the occurrence of thromboembolic events (within one week of delivery).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women candidate for LSCS.
* Age: 20-40 years old.
* Full term pregnancies (> 37 weeks confirmed by the 1st day of the LMP or 1st trimesteric ultrasound scan).
* Singleton or twin pregnancies.
* Maternal Anemia (hemoglobin < 9.9 g%)
* Maternal medical disorders (e.g. cardiac, renal, and hepatic diseases, Thromboembolic disorders or coagulopathies).
* High risk case for obstetric hemorrhage (e.g. peripartum hemorrhage, accidental hemorrhage, placenta previa, previous history of uterine atony or postpartum hemorrhage).
* CS under spinal anesthesia.

Exclusion Criteria:

* Fetal death (IUFD).
* Fetal anomalies or IUGR (estimated fetal weight below the 5th centile)
* Women attending for emergency CS.
* More than 2 previous CS procedures.
* Prolonged procedure (more than 2 hours from skin incision to skin closure).
* History of prostaglandin or Tranexamic acid allergy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 345 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
o compare the estimated blood loss (EBL) during cesarean delivery among the three groups | Intraoperative and within the first 24 hours postoperative.
  Estimated Blood Loss (EBL) will be evaluated as follows:
  A. The number of operative towels used. B. The difference of weight of operative towels (before and after cs) plus the amount of blood in suction unit (we will calculate 1 gram of weight difference equal to 1 ml blood loss).
  C. EBL calculation according to the following formula:
  EBL= EBV x [(Preoperative hematocrit- Postoperative hematocrit)/ Postoperative hematocrit]

SECONDARY OUTCOMES:
The Use of additional ecbolics denoting uterine atony | within 24 hours postpartum
  5 IU intravenous bolus oxytocin and 1mL [0.2 mg] intramuscular ergometrine with or without 600 microgram rectal misoprostol postoperatively).
The occurrence of Excessive blood loss will be documented | within the first 24 hours postoperatively
  Excessive blood loss (> 1000 mL) and the need for blood transfusion will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Moutaz Elsherbini, MD, Principal Investigator — assistant professor
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawoud M, Al-Husseiny M, Helal O, Elsherbini M, Abdel-Rasheed M, Sediek M. Intravenous tranexamic acid vs. sublingual misoprostol in high-risk women for postpartum haemorrhage following cesarean delivery; a randomised clinical trial. BMC Pregnancy Childbirth. 2023 Aug 25;23(1):611. doi: 10.1186/s12884-023-05935-5. PMID 37626292